CLINICAL TRIAL: NCT01350414
Title: AIR2 Extension Study to Demonstrate Longer-term (> 1 Year) Durability of Effectiveness
Acronym: PAS1
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 10-01
Record Dates: First submitted 2010-10-28; First posted 2011-05-09 (Estimated); Results first posted 2016-09-26 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Alair Group: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02, NCT00231114)
  Interventions: Device: Bronchial Thermoplasty with the Alair System

INTERVENTIONS:
Device: Bronchial Thermoplasty with the Alair System — Bronchial Thermoplasty with the Alair System

SUMMARY:
The objective of this study is to evaluate durability of effectiveness (beyond one year) of the Alair System in patients with severe persistent asthma. The study will consist of Alair-group subjects who are currently in the follow-up phase (out to 5 years) of the AIR2 Trial (Protocol #04-02, clinicaltrials.gov number NCT00231114).

Durability of the treatment effect will be evaluated by comparing the proportion of subjects who experience severe exacerbations during the first year after Alair treatment with the proportion of subjects who experience severe exacerbations during subsequent 12 month periods out to 5 years.

All Alair group subjects in the AIR2 Trial are being followed out to 5 years as per the AIR2 Trial protocol. The data that are to be used to determine durability of effectiveness as described in the present protocol (Protocol #10-01) are being collected under the existing AIR2 Trial protocol (Protocol # 04-02).

Study Hypothesis: An empirical demonstration of the durability of the treatment effect will be used to show that the proportion of subjects experiencing severe exacerbations for the first year compared with the proportions of subjects experiencing severe exacerbations in subsequent years do not get substantially worse.

The primary statistical objective is to demonstrate that the proportion of subjects who experience severe exacerbations in the subsequent 12-month follow-up (for Year 2, Year 3, Year 4 and Year 5 [in 12-month periods]) is not statistically worse when compared with the proportion of first 12-months, which begins 6-weeks after the last Alair treatment. This objective will be met if the upper 95% confidence limit of the difference in proportions (i.e., the subsequent 12-month proportion minus the first 12-month proportion) is less than 20%.

DETAILED DESCRIPTION:
This will be an open-label, single arm study designed to demonstrate the durability of effectiveness (beyond one year) of the Alair System in patients with severe persistent asthma.

Durability of treatment effect will be evaluated by comparison of the proportion of subjects experiencing severe exacerbations during the first year after the Alair treatment to subsequent 12-month periods out to 5 years.

The 12-month periods will begin 6 weeks post-last Alair bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All Alair group subjects who have participated in the AIR2 Trial (NCT00231114) and were not lost to follow-up at the end of the 12 month premarket visit, and those who are willing to comply with the study protocol and routine visits for the duration of the study will be included in the post-approval study

Exclusion Criteria:

* None.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Alair group subjects who have participated in the AIR2 Trial (NCT00231114) and were not lost to follow-up at the end of the 12 month premarket visit, and those who are willing to comply with the study protocol and routine visits for the duration of the study will be included in the post-approval study.
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2005-10; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder S Shargill, PhD, Study Director — Asthmatx, Inc.

REFERENCES:
- [Background] Castro M, Rubin AS, Laviolette M, Fiterman J, De Andrade Lima M, Shah PL, Fiss E, Olivenstein R, Thomson NC, Niven RM, Pavord ID, Simoff M, Duhamel DR, McEvoy C, Barbers R, Ten Hacken NH, Wechsler ME, Holmes M, Phillips MJ, Erzurum S, Lunn W, Israel E, Jarjour N, Kraft M, Shargill NS, Quiring J, Berry SM, Cox G; AIR2 Trial Study Group. Effectiveness and safety of bronchial thermoplasty in the treatment of severe asthma: a multicenter, randomized, double-blind, sham-controlled clinical trial. Am J Respir Crit Care Med. 2010 Jan 15;181(2):116-24. doi: 10.1164/rccm.200903-0354OC. Epub 2009 Oct 8. PMID 19815809
- [Result] Wechsler ME, Laviolette M, Rubin AS, Fiterman J, Lapa e Silva JR, Shah PL, Fiss E, Olivenstein R, Thomson NC, Niven RM, Pavord ID, Simoff M, Hales JB, McEvoy C, Slebos DJ, Holmes M, Phillips MJ, Erzurum SC, Hanania NA, Sumino K, Kraft M, Cox G, Sterman DH, Hogarth K, Kline JN, Mansur AH, Louie BE, Leeds WM, Barbers RG, Austin JH, Shargill NS, Quiring J, Armstrong B, Castro M; Asthma Intervention Research 2 Trial Study Group. Bronchial thermoplasty: Long-term safety and effectiveness in patients with severe persistent asthma. J Allergy Clin Immunol. 2013 Dec;132(6):1295-302. doi: 10.1016/j.jaci.2013.08.009. Epub 2013 Aug 30. PMID 23998657

RESULTS

PARTICIPANT FLOW:
Groups:
- Alair Group: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02)
  Bronchial Thermoplasty with the Alair System: Bronchial Thermoplasty with the Alair System
Period: Overall Study
Arm/Group | Alair Group
Started | 181
Year 2 | 165
Year 3 | 162
Year 4 | 159
Year 5 | 162
Completed | 162
Not Completed | 19
Not completed — Lost to Follow-up | 13
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 2

BASELINE CHARACTERISTICS:
Population: AIR2 Extension Subjects Completing Follow-up at Year 1
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.8 (11.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 102
  Male | 79
Region of Enrollment [Number; unit: participants]
  Brazil | 54
  Canada | 34
  United States | 54
  Australia | 7
  United Kingdom | 27
  Netherlands | 5
Height (cm) [Mean (Standard Deviation); unit: cm] | 166.8 (8.94)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 81.9 (17.95)
ICS Dose (Inhaled Corticosteroid dose) [Mean (Standard Deviation); unit: mcg/day (micrograms/day)] | 1943.9 (722.39)
LABA Dose (Long-acting Beta Agonists) [Mean (Standard Deviation); unit: mcg/day] | 119.2 (45.64)
OCS Dose (Oral corticosteroids) [Mean (Standard Deviation); unit: mg/day] — This measure includes only 7 participants using OCS at baseline.
  mg/day | 6.4 (1.97)
Asthma Quality of Life Questionnaire (AQLQ) Score [Mean (Standard Deviation); unit: Scores on a scale] — There are 32 questions in the AQLQ and they are in 4 domains (symptoms, activity limitation, emotional function and environmental stimuli). Patients are asked to think about how they have been during the previous two weeks and to respond to each of the 32 questions on a 7-point scale (7 = not impaired at all - 1 = severely impaired). The overall AQLQ score is the mean of all 32 responses and the individual domain scores are the means of the items in those domains.
  Scores on a scale | 4.32 (1.15)
Pre-Bronchodilator FEV1 (Forced Expiratory Volume in 1 second) [Mean (Standard Deviation); unit: % predicted] | 77.8 (15.67)
Post-Bronchodilator FEV1 (Forced Expiratory Volume in 1 second) [Mean (Standard Deviation); unit: % predicted] | 86 (15.65)
amPEF (Peak Expiratory Flow) [Mean (Standard Deviation); unit: L/min (liters per minute)] | 383.4 (104.65)

OUTCOME MEASURES:

1. Primary Outcome: Severe Exacerbations
Description: The primary endpoint will be the proportion of subjects experiencing severe exacerbations during the first year after the Alair treatment compared to subsequent 12-month periods out to 5 years. This objective will be met if the upper 95% confidence limit of the difference in proportions (i.e., the subsequent 12-month proportion minus the first 12-month proportion) is less than 20%.
  Severe exacerbation is defined as treatment with oral or intravenous corticosteroids, OR a doubling of the baseline inhaled corticosteroid dose for at least 3 days, OR any temporary increase in the dosage of oral corticosteroids for a subject taking maintenance oral corticosteroids at entry into the AIR2 Trial (Protocol #04-02).
Time Frame: 12 month periods out to 5 Years
Population: Number of Subjects Completing Follow-up. 181 subjects completed 12 month follow-up; 165 subjects completed Year 2 follow-up; 162 subjects completed Year 3 follow-up; 159 subjects completed Year 4 follow-up; and 162 subjects completed Year 5 follow-up.
Measure: Number (95% Confidence Interval); unit: Percentage subjects severe exacerbations
Groups:
- Alair Group: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol number 04-02, NCT00231114).
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Percentage subjects severe exacerbations
  Year 1 | 30.9 [24.2 to 37.7]
  Year 2 | 23.6 [17.2 to 30.1]
  Year 3 | 34 [26.7 to 41.2]
  Year 4 | 36.5 [29 to 44]
  Year 5 | 21.6 [15.3 to 27.9]

2. Secondary Outcome: Severe Exacerbations
Description: Number of severe exacerbations per subject per year. Severe exacerbation is defined as treatment with oral or intravenous corticosteroids, OR a doubling of the baseline inhaled corticosteroid dose for at least 3 days, OR any temporary increase in the dosage of oral corticosteroids for a subject taking maintenance oral corticosteroids at entry into the AIR2 Trial (Protocol #04-02).
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of events/Number of subjects/Year
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Number of events/Number of subjects/Year
  Year 1 | 0.486 [0.385 to 0.614]
  Year 2 | 0.406 [0.311 to 0.531]
  Year 3 | 0.549 [0.435 to 0.693]
  Year 4 | 0.560 [0.444 to 0.706]
  Year 5 | 0.309 [0.226 to 0.421]

3. Secondary Outcome: Respiratory Adverse Events
Description: Number of respiratory adverse events per subject per year. A respiratory adverse event is defined as any sign, symptom, illness, clinically significant abnormal laboratory value, or other adverse medical event associated with the "Respiratory System" that appears or worsens in a subject during a clinical study, regardless of whether or not it is considered related to the procedure used as part of the protocol.
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of events/number of subject/Year
Groups:
- Alair Group: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02).
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Number of events/number of subject/Year
  Year 1 | 2.022 [1.764 to 2.318]
  Year 2 | 1.218 [1.013 to 1.465]
  Year 3 | 1.247 [1.037 to 1.499]
  Year 4 | 1.176 [0.971 to 1.424]
  Year 5 | 0.778 [0.616 to 0.982]

4. Secondary Outcome: Respiratory Adverse Events
Description: Proportion of subjects experiencing one or more respiratory adverse event in each of the years 1 through 5 following the Alair treatment. A respiratory adverse event is defined as any sign, symptom, illness, clinically significant abnormal laboratory value, or other adverse medical event associated with the "Respiratory System" that appears or worsens in a subject during a clinical study, regardless of whether or not it is considered related to the procedure used as part of the protocol.
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage subjects with respiratory AE
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Percentage subjects with respiratory AE
  Year 1 | 72.9 [66.5 to 79.4]
  Year 2 | 58.8 [51.3 to 66.3]
  Year 3 | 58 [50.4 to 65.6]
  Year 4 | 54.7 [47 to 62.5]
  Year 5 | 47.5 [39.8 to 55.2]

5. Secondary Outcome: Emergency Room Visits for Respiratory Symptoms
Description: Proportion of Subjects with Emergency Room Visits for Respiratory Symptoms
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage subjects ER respir. symptoms
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Percentage subjects ER respir. symptoms
  Year 1 | 5 [1.8 to 8.1]
  Year 2 | 6.7 [2.9 to 10.5]
  Year 3 | 8 [3.8 to 12.2]
  Year 4 | 6.9 [3 to 10.9]
  Year 5 | 5.6 [2 to 9.1]

6. Secondary Outcome: Emergency Room (ER) Visits for Respiratory Symptoms
Description: Number of Emergency Room Visits for Respiratory Symptoms per subject per year.
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of events/subject/year
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Number of events/subject/year
  Year 1 | 0.072 [0.048 to 0.107]
  Year 2 | 0.085 [0.058 to 0.124]
  Year 3 | 0.136 [0.100 to 0.184]
  Year 4 | 0.094 [0.065 to 0.136]
  Year 5 | 0.068 [0.044 to 0.104]

7. Secondary Outcome: Hospitalizations for Respiratory Symptoms
Description: Proportion of subjects with hospitalizations for respiratory symptoms.
Time Frame: 12 Month periods out to 5 Years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of subjects hospitalized
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Percentage of subjects hospitalized
  Year 1 | 3.3 [0.7 to 5.9]
  Year 2 | 4.2 [1.2 to 7.3]
  Year 3 | 6.2 [2.5 to 9.9]
  Year 4 | 5.7 [2.1 to 9.3]
  Year 5 | 1.9 [0.0 to 3.9]

8. Secondary Outcome: Hospitalizations for Respiratory Symptoms
Description: Number of Hospitalizations for Respiratory Symptoms per subject per year.
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Number of events/subjects/year
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Number of events/subjects/year
  Year 1 | 0.039 [0.025 to 0.060]
  Year 2 | 0.061 [0.042 to 0.087]
  Year 3 | 0.068 [0.048 to 0.096]
  Year 4 | 0.075 [0.054 to 0.105]
  Year 5 | 0.025 [0.014 to 0.044]

9. Secondary Outcome: Pre-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: Pre-Bronchodilator FEV1 (% Predicted) percentage changes from Baseline to the Year 1, Year 2, Year 3, Year 4, and Year 5.
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change from Baseline
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Percentage of change from Baseline
  Year 1 | -1.4 (14.82)
  Year 2 | -4.6 (15.36)
  Year 3 | -2.7 (15.33)
  Year 4 | -1.2 (14.60)
  Year 5 | -1.2 (16.33)

10. Secondary Outcome: Post-Bronchodilator Forced Expiratory Volume in 1 Second (FEV1)
Description: Post-Bronchodilator FEV1 (% Predicted) percentage changes from Baseline to the Year 1, Year 2, Year 3, Year 4, and Year 5.
Time Frame: 12 Month periods out to 5 years
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of change from Baseline
Arm/Group | Alair Group
Number analyzed (Participants) | 181
Percentage of change from Baseline
  Year 1 | -2.8 (10.67)
  Year 2 | -5.4 (11.51)
  Year 3 | -4 (12.88)
  Year 4 | -3.7 (11.65)
  Year 5 | -3.8 (11.95)

ADVERSE EVENTS:
Time Frame: 12 months out to 5 years
Description: In previous outcome analysis and in the participant flow, the denominator was based on the number of subjects that completed the corresponding annual visit. For Adverse Events the denominator was based on all the subjects that entered that period regardless of whether they completed the annual visit or not for that period.
Groups:
- Year 1: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02).
  Year 1 is defined as 365 days from the treatment period (6 weeks after the last bronchoscopy). All subjects were considered in the analysis regardless of whether they have completed the Year 1 annual visit or not.
- Year 2: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02).
  Year 2 is defined as 366 to 730 days after the treatment period. All subjects were considered in the analysis regardless of whether they have completed the Year 2 annual visit or not.
- Year 3: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02).
  Year 3 is defined as 731 to 1095 days after the treatment period. All subjects were considered in the analysis regardless of whether they have completed the Year 3 annual visit or not.
- Year 4: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02).
  Year 4 is defined as 1096 to 1460 days after the treatment period. All subjects were considered in the analysis regardless of whether they have completed the Year 4 annual visit or not.
- Year 5: Subjects who underwent treatment with the Alair System in the AIR2 Trial (Protocol No. 04-02).
  Year 5 is defined as 1461 days to 1826 days after the treatment period. All subjects were considered in the analysis regardless of whether they have completed the Year 5 annual visit or not.
Arm/Group | Year 1 | Year 2 | Year 3 | Year 4 | Year 5
Serious Adverse Events (participants affected / at risk) | 5/187 | 8/168 | 10/163 | 9/163 | 3/162
Other Adverse Events (participants affected / at risk) | 112/187 | 89/168 | 81/163 | 77/163 | 61/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 1 (N=187) | Year 2 (N=168) | Year 3 (N=163) | Year 4 (N=163) | Year 5 (N=162)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-respiratory
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Addison's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Anorectal disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Non-respiratory
Abscess limb (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-respiratory
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Infective tenosynovitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Osteomyelitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Perianal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Viral labyrinthitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Non-respiratory
Traumatic brain injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Obesity (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Non-respiratory
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Non-respiratory
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (8) | 7 (8) | 6 (9) | 2 (3) — Respiratory
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Respiratory
Chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Lobar pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Respiratory
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) — Respiratory
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Respiratory
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Non-respiratory
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Year 1 (N=187) | Year 2 (N=168) | Year 3 (N=163) | Year 4 (N=163) | Year 5 (N=162)
Asthma (Respiratory, thoracic and mediastinal disorders) | 52 (87) | 47 (77) | 48 (82) | 51 (81) | 40 (52) — Respiratory
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 14 (18) | 12 (14) | 8 (11) | 6 (7) | 5 (6) — Respiratory
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 9 (15) | 11 (14) | 15 (20) | 6 (7) — Respiratory
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 21 (27) | 9 (10) | 6 (7) | 6 (6) | 1 (1) — Respiratory
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 12 (16) | 16 (17) | 11 (14) | 9 (10) | 6 (7) — Respiratory
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 57 (81) | 24 (29) | 24 (25) | 23 (28) | 18 (23) — Respiratory
Viral upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 6 (6) | 1 (1) | 1 (1) | 3 (3) — Respiratory

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less